CLINICAL TRIAL: NCT04039854
Title: Comparison Between Propofol and Inhalational Anaesthetic Agents on Cardiovascular Outcomes Following Cardiac Surgery - a Randomised Controlled Feasibility Trial
Brief Title: Comparison Between Propofol and Inhalational Anaesthetic Agents on Cardiovascular Outcomes Following Cardiac Surgery
Acronym: COPIA
Status: Unknown | Phase: Phase 4 | Type: Interventional
Last Known Status: Recruiting
Sponsor: King's College Hospital NHS Trust (Other)
Collaborators: London School of Hygiene and Tropical Medicine (Other); Guy's and St Thomas' NHS Foundation Trust (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: KCH-PRO:19/001; 2019-000171-16 (EudraCT Number); 216646 (Other: IRAS ID)
Record Dates: First submitted 2019-06-07; First posted 2019-07-31 (Actual); Last update posted 2021-02-24 (Actual); Status verified 2021-02

CONDITIONS: Coronary Heart Disease; Cardiovascular Diseases
Keywords: Anaesthesia; Coronary Artery Bypass Surgery; Cardioprotection
MeSH Terms: conditions — Coronary Disease; Cardiovascular Diseases | interventions — Isoflurane; Sevoflurane; Desflurane; Propofol

STUDY DESIGN:
Who Masked: Participant
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (2):
- Volatile anaesthetics arm (Active Comparator): Patients randomised to receive volatile anaesthetics will receive either isoflurane, sevoflurane or desflurane during the surgical procedure.
  Interventions: Drug: Isoflurane, Sevoflurane or Desflurane
- Propofol anaesthetics arm (Active Comparator): Patients randomised to receive propofol will not receive any volatile anaesthetics during the surgical procedure.
  Interventions: Drug: Propofol

INTERVENTIONS:
Drug: Isoflurane, Sevoflurane or Desflurane — The volatile anaesthetic agent will be administered via inhalation, i.e. ventilation through alveolar membrane in lungs) during the maintenance of anaesthesia. During CPB the volatile anaesthetic agent will be administered through the oxygenator oxygen inflow of the CPB machine.
  The maintenance dose of the volatile anaesthetic agent will be titrated to doses deemed necessary in order to provide sufficient depth of anaesthesia and blood pressure.
  The administration of the volatile anaesthetic agent will be started after induction of anaesthesia and it will be ended at the end of surgery, before the patient is transferred to the CCU.
  Arms: Volatile anaesthetics arm
Drug: Propofol — Patients will receive propofol only during the surgical procedure. The maintenance dose of the propofol infusion will be titrated to doses deemed necessary in order to provide sufficient depth of anaesthesia (titrated to a depth of anaesthesia with BIS 30-60) and mean arterial pressure (MAP) of 50-80mmHg by the treating anaesthetist.
  Arms: Propofol anaesthetics arm

SUMMARY:
The objective of this research proposal is to find out whether comparing the two different anaesthetic maintenance techniques (Propofol vs volatile anaesthetics) in adult patients undergoing heart surgery is practical for the anaesthetist treating the patients and whether it is feasible for the research team to recruit patients and follow them up after the operation.

DETAILED DESCRIPTION:
All patients undergoing heart bypass surgery are given anaesthetics during the operation. There are two types of anaesthetic commonly given to patients undergoing heart bypass surgery.

Propofol is an anaesthetic that is delivered into the patient's vein. Other anaesthetics which are inhaled include Isoflurane, Sevoflurane and Desflurane and these are called volatile anaesthetics. Preliminary studies over the past ten years suggests that maintenance of general anaesthesia using only volatile anaesthetics has the potential to improve health outcomes after bypass surgery, when compared with propofol.

Volatile anaesthetics have been shown to protect the heart, the kidneys and the brain, however results of studies have been inconclusive. Currently both volatile anaesthetics and propofol are used equally in clinical practice in the UK.

ELIGIBILITY:
Inclusion Criteria:

* Patients (male and female) aged 18 years and above
* Written informed consent to participate
* Patients undergoing Coronary Artery Bypass Graft (CABG) surgery on Cardiopulmonary bypass (CPB) with or without valve surgery
* Additive European System for Cardiac Operative Risk Evaluation (EuroSCORE) of 5 or higher

Exclusion Criteria:

* Pregnant or lactating women
* Allergy to propofol
* Previous diagnosis or suspected malignant hyperthermia
* Patients with a known sensitivity to any of the IMPs or other halogenated anaesthetics
* Concomitant therapy with glibenclamide or nicorandil (medications that may interfere with preconditioning)
* Inclusion in another clinical trial of an investigational medicinal product within the last 3 months.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 50 (Estimated)
Dates: Start 2019-11-20 (Actual); Primary Completion 2021-11-30 (Estimated); Study Completion 2022-01-31 (Estimated)

PRIMARY OUTCOMES:
Recruitment rate | Collected over the recruitment period of 10 months
  To identify whether it is feasible to recruit up to 50 patients across 2 tertiary cardiac surgery centres within approximately 10 months.
To identify barriers to recruitment. | Collected over the recruitment period of 10 months
  This data will be completed on a screening log.

SECONDARY OUTCOMES:
Feasibility of maintaining follow-up rates of over 95% | Collected over the recruitment period of 10 months
  This data will be gathered in the trial database.
Assessment of effectiveness of patient identification and screening processes | Collected over the recruitment period of 10 months
  To record the number of patients screened and potentially eligible for the trial at the two tertiary cardiac surgery centres within a period of 10 months. This data will be gathered on the screening log.
To investigate whether it is feasible to recruit at least 10% of all potentially eligible patients at the two tertiary cardiac surgery centres within a period of 10 months. | Collected over the recruitment period of 10 months
  This data will be gathered on screening logs and in the randomisation system.
To investigate whether it is feasible to maintain routine data collection and follow up rates greater than 90% over the trial period. | Collected over the full trial period of 24 months
  This data will be gathered in the randomisation site and trial database.
To investigate whether it is feasible to achieve 95% data collection of Low Cardiac Output Syndrome for the full trial over the trial period. | Collected over the full trial period of 24 months
  This data will be gathered in the trial database.
To investigate whether it is feasible to achieve 95% data collection of Myocardial injury, assessed by ischaemic serum markers: hsTnT, MyC, for the full trial over the trial period. | Preop, 6 hrs after arrival in CCU, and postop day 1 and 2. Collected over the full trial period of 24 months
  This data will be gathered in the trial database.
To investigate whether it is feasible to achieve 90% data collection of MACCE (stroke, non-fatal myocardial infarction, death from any cause) for the full trial over the trial period. | Data collected at 30 days post op.
  This data will be gathered in the trial database.
To investigate whether it is feasible to achieve 90% data collection of Cardiac related mortality at 30 days for the full trial over the trial period. | Data collected at 30 days post op.
  This data will be gathered in the trial database.
To investigate whether it is feasible to achieve 90% data collection of Postoperative in hospital atrial fibrillation requiring treatment for the full trial over the trial period. | Data collected at 30 days post op.
  This data will be gathered in the trial database.
To investigate whether it is feasible to achieve 90% data collection of Acute Kidney Injury (according to Kidney Disease: Improving Global Outcomes guidelines) for the full trial over the trial period. | Data collected at 30 days post op.
  AKI will be confirmed by a 1.5 - 1.9 increase of serum creatinine from baseline or an absolute value rise of creatine greater than 0.3mg/dl (27mmol/L) from baseline. This data will be gathered in the trial database.
To investigate whether it is feasible to achieve 90% data collection of In-hospital postoperative delirium (assessed by the confusion assessment method) for the full trial over the trial period. | Data collected at 30 days post op.
  This data will be gathered in the trial database.
To investigate whether it is feasible to achieve 90% data collection of Respiratory complications needing prolonged ventilation (>24 hours) for the full trial over the trial period. | Data collected at 30 days post op.
  This data will be gathered in the trial database.
To investigate whether it is feasible to achieve 90% data collection of Length of stay in the critical care unit (CCU) for the full trial over the trial period. | Data collected at 30 days post op.
  This data will be gathered in the trial database.
To investigate whether it is feasible to achieve 90% data collection of Length of hospital stay for the full trial over the trial period. | Data collected at 30 days post op.
  This data will be gathered in the trial database.
To investigate whether it is feasible to achieve 90% data collection of WHO Disability Assessment Schedule (WHODAS) for the full trial over the trial period. | Data collected at 30 days post op.
  This data will be gathered in the trial database.
To investigate whether it is feasible to achieve 90% data collection of Quality of Life Questionnaire (Euroqol, EQ-5D-5L) for the full trial over the trial period. | Data collected at Baseline and 30 days postoperative
  This data will be gathered in the trial database.
To investigate whether it is feasible to achieve 90% data collection of Days alive and at home for the full trial over the trial period. | Data collected at 30 days postoperative
  This data will be gathered in the trial database.

CONTACTS AND LOCATIONS:
Overall Officials: Dr Gudrun Kunst, Principal Investigator — King's College Hospital NHS Trust
Locations (2):
- United Kingdom (2):
  - St Thomas' Hospital, London
  - Kings College Hospital NHS Foundation Trust, London

IPD SHARING:
Plan to Share IPD: Yes
Anonymous participant data may be shared with other researchers

REFERENCES:
- [Derived] Milne B, John M, Evans R, Robertson S, O Scanaill P, Murphy GJ, Landoni G, Marber M, Clayton T, Kunst G. Comparison between propofol and total inhalational anaesthesia on cardiovascular outcomes following on-pump cardiac surgery in higher-risk patients: a randomised controlled pilot and feasibility study. Open Heart. 2024 May 9;11(1):e002630. doi: 10.1136/openhrt-2024-002630. PMID 38724266